CLINICAL TRIAL: NCT00786149
Title: Improving Varenicline Adherence and Outcomes in Homeless Smokers
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0708M14444; HL081522; NIH-522
Record Dates: First submitted 2008-11-05; First posted 2008-11-06 (Estimated); Last update posted 2014-09-03 (Estimated); Status verified 2014-09

CONDITIONS: Tobacco Use Cessation
Keywords: Underserved populations; Homelessness; Nicotine replacement therapy; Counseling; Cancer Prevention and control
MeSH Terms: conditions — Tobacco Use Cessation | interventions — Varenicline; Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Participants will receive NRT and Motivational Interviewing counseling
  Interventions: Other: Varenicline plus Motivational Interviewing counseling
- 2 (Active Comparator): Varenicline plus brief advice
  Interventions: Other: Varenicline without counseling

INTERVENTIONS:
Other: Varenicline plus Motivational Interviewing counseling — Motivational Interviewing; 8 weeks of counseling
  Other Names: Chantix
  Arms: 1
Other: Varenicline without counseling — Brief advice, one time during initial session
  Other Names: Chantix
  Arms: 2

SUMMARY:
the purpose of the study is to see if varenicline in combination with motivational counseling helps homeless cigarette smokers quit smoking.

DETAILED DESCRIPTION:
Despite significant declines in cigarette smoking rates among adults in the United States in the last few decades, smoking rates remain high among poor and underserved populations. One underserved group is the 4 million homeless persons in the US among whom cigarette smoking rate is an alarming 70% or more; these rates are 3 times higher than national average. Two of the three leading causes of death among homeless persons, heart disease and cancer are tobacco related.2, 3 Despite very high smoking prevalence and disease burden in this population smoking cessation research have not been extended to the homeless. Recent studies including data from our research team show a considerable degree of readiness to quit smoking by homeless smokers and that nicotine replacement therapy (NRT) plus counseling show promise. However, homeless persons face many challenges that may constitute barriers for them to adhere to smoking cessation treatments even if such treatments have been proven effective in the general population. In order to reduce smoking-related health disparities within this underserved population, it is critical that cessation interventions including strategies to improve treatment adherence be developed to include homeless smokers. The primary aim of this study is to assess the effects of adherence-focused motivational interviewing (MI) to help homeless persons quit smoking.

Recruitment and retention will be enhanced by use of bus passes for transportation, debit cards, attractive intervention materials, collaboration with homeless shelters, and advice from a community advisory board. If successful, this study will provide a model for how to overcome barriers to cancer prevention services among homeless persons. It will also provide the impetus for policy changes directed at increasing homeless persons' access to smoking cessation pharmacotherapy and treatment.

ELIGIBILITY:
Inclusion Criteria:

* currently homeless
* smoke 5 or more cigarettes per day
* smoked 100 cigarettes in lifetime
* aged 18 years or older

Exclusion Criteria:

* unstable mental illness
* pregnancy
* current history of psychoactive or alcohol dependence or psychotic disorder
* cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 428 (Actual)
Dates: Start 2007-09; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
7-day point prevalence abstinence from smoking | 6 months after enrollment

SECONDARY OUTCOMES:
Adherence to treatment | 12 weeks and 6 months after enrollment
Moderating effects of psychiatric co-morbidities and other substance abuse on treatment | 6 months after enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Kolawole S Okuyemi, MD,MPH, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Theodoulou A, Fanshawe TR, Leavens E, Theodoulou E, Wu AD, Heath L, Stewart C, Nollen N, Ahluwalia JS, Butler AR, Hajizadeh A, Thomas J, Lindson N, Hartmann-Boyce J. Differences in the effectiveness of individual-level smoking cessation interventions by socioeconomic status. Cochrane Database Syst Rev. 2025 Jan 27;1(1):CD015120. doi: 10.1002/14651858.CD015120.pub2. PMID 39868569
- [Derived] Ojo-Fati O, Joseph AM, Ig-Izevbekhai J, Thomas JL, Everson-Rose SA, Pratt R, Raymond N, Cooney NL, Luo X, Okuyemi KS. Practical issues regarding implementing a randomized clinical trial in a homeless population: strategies and lessons learned. Trials. 2017 Jul 5;18(1):305. doi: 10.1186/s13063-017-2046-9. PMID 28679430
- [Derived] Ojo-Fati O, Thomas JL, Vogel RI, Ogedegbe O, Jean-Louis G, Okuyemi KS. Predictors of Adherence to Nicotine Replacement Therapy (Nicotine Patch) Among Homeless Persons Enrolled in a Randomized Controlled Trial Targeting Smoking Cessation. J Fam Med. 2016;3(7):1079. Epub 2016 Sep 6. PMID 28580456
- [Derived] Goldade K, Whembolua GL, Thomas J, Eischen S, Guo H, Connett J, Des Jarlais D, Resnicow K, Gelberg L, Owen G, Grant J, Ahluwalia JS, Okuyemi KS. Designing a smoking cessation intervention for the unique needs of homeless persons: a community-based randomized clinical trial. Clin Trials. 2011 Dec;8(6):744-54. doi: 10.1177/1740774511423947. PMID 22167112